CLINICAL TRIAL: NCT06135571
Title: Real World Registry Study on the No.253 Lymph Node Metastasis Patterns in Left-Sided Colon and Rectal Cancer
Brief Title: Study on the No.253 Lymph Node Metastasis Patterns in Left-Sided Colon and Rectal Cancer
Status: Recruiting | Type: Observational
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Collaborators: Peking Union Medical College Hospital (Other); Peking University Cancer Hospital & Institute (Other); China-Japan Friendship Hospital (Other); Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, QIAN LIU, Professor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Other Study IDs: NCC4280
Record Dates: First submitted 2023-11-12; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Colorectal Cancer; Lymph Node Metastasis
Keywords: Left-sided colorectal cancer; Lymph node dissection; No.253 lymph node
MeSH Terms: conditions — Colorectal Neoplasms; Lymphatic Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort of left-sided colorectal cancer: Patients underwent curative surgery with dissection of No.253 Lymph node
  Interventions: Procedure: Laparoscopic colorectal surgery

INTERVENTIONS:
Procedure: Laparoscopic colorectal surgery — Patients underwent laparoscopic left colectomy, sigmoid resection or rectal surgery according to the location of tumor.

SUMMARY:
The goal of this observational study is to learn about the the pattern of metastasis of the No.253 lymph node in colorectal cancer. The main questions it aims to answer are: 1. What are the risk factors for metastasis to the No.253 lymph node? 2.What is the prognosis for patients with metastasis to the No.253 lymph node? Patients with descending colon cancer, sigmoid colon cancer, and rectal cancer who undergo curative surgery with dissection of the No.253 lymph node are included in this study

DETAILED DESCRIPTION:
The No. 253 lymph node (also named as apical lymph node of inferior mesenteric artery), as the third station in the inferior mesenteric artery lymphatic system, plays a vital role in the lymphatic circulation of the descending colon, sigmoid colon, and rectum. They serve as the last barrier for tumor metastasis from regional to distant sites. The definition of the range of the No.253 lymph node primarily follows the Japanese Colorectal Cancer Treatment Guidelines: the medial boundary is the segment from the root of the inferior mesenteric artery to the origin of the left colic artery, the caudal boundary is from the origin of the left colic artery to the intersection with the inferior mesenteric vein, the lateral boundary is the outer margin of the inferior mesenteric vein, and the cranial boundary is from the horizontal section of the duodenum to the beginning of the jejunum. However, the pattern of metastasis of the No.253 lymph node in colorectal cancer remains unclear, with most studies being retrospective and showing significant differences in results. Therefore, the investigator plans to be the first internationally to carry out this retrospective, registry-based study to determine the metastasis pattern to the No. 253 lymph node in colorectal cancer. This will provide definitive clinical evidence for D3 lymph node dissection in colorectal surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-75 years;
2. Underwent laparoscopic left hemicolectomy, sigmoid colectomy, or rectal cancer radical surgery.
3. Postoperative pathology confirmed as adenocarcinoma.
4. No evidence of distant metastasis.

Exclusion Criteria:

1. Previous history of malignant colorectal tumors.
2. Patients who have undergone multiple abdominal-pelvic surgeries.
3. Patients undergoing emergency surgery due to complications such as intestinal obstruction, intestinal perforation, or intestinal bleeding.
4. Surgery did not achieve R0 resection.
5. Patients with concurrent other malignant tumors or multiple primary colorectal cancers.
6. Patients unwilling to sign an informed consent or follow the study protocol for follow-up.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with left-sided colorectal cancer (left colon cancer, sigmoid cancer, rectal cancer) underwent laparoscopic surgery with dissection of No.253 lymph node.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Metastatic rate of No.253 lymph node | About 10 days after surgery
  Pathologically confirmed tumor cell infiltration in the No.253 lymph node

SECONDARY OUTCOMES:
Number of harvested lymph nodes | About 10 days after surgery
  Total number of lymph nodes dissected in the pathology report
Incidence of postoperative complications | 30 days after surgery
  The proportion of short-term complications occurring within 30 days post-surgery
5-year local recurrence rate | 5 years after surgery
  Local recurrence refers to the return of cancer in the same area where it originally developed, typically after treatment has been completed.
5-year disease free survival rate | 5 years after surgery
  Disease free survival refers to the length of time after primary treatment during which a patient survives without any signs or symptoms of the cancer.
5-year overall survival rate | 5 years after surgery
  Overall survival refers to the length of time from the primary treatment that patients are still alive.

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Chinese PLA General Hospital, Beijing, Beijng

IPD SHARING:
Plan to Share IPD: No